CLINICAL TRIAL: NCT04552353
Title: A Randomized, Single-dose, Two-way Crossover Study to Evaluate Bioequivalence of Two Formulations of Voriconazole(200mg/Vial) After Intravenous Infusion of 200mg Voriconazole in Healthy Volunteers Under Fasting Conditions.
Brief Title: Evaluate Bioequivalence of Voriconazole(200mg/Vial) .
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YSP-RKH3003-01
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Antimycotic for Systematic Use
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaway Lyo-Injection (Experimental): Voriconazole, 200 mg/vial
  Interventions: Drug: Vaway
- Vfend Lyo-Injection (Active Comparator): Voriconazole, 200 mg/vial
  Interventions: Drug: Vaway

INTERVENTIONS:
Drug: Vaway — Drug: Voriconazole. Pharmacokinetic study under fasting conditions
  Other Names: Vfend

SUMMARY:
A Randomized, Single-dose, Two-way Crossover Study to Evaluate Bioequivalence of Two Formulations of Voriconazole(200mg/Vial) After Intravenous Infusion of 200mg Voriconazole in Healthy Volunteers Under Fasting Conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subjects between 20-45 years of age (inclusive) at the screening visit.
2. Body weight within 80-120% of ideal body weight but not less than 45kg at the screening visit.

   * Ideal body weight (kg) = [height (cm) - 80] ´ 0.7 for male subjects
   * Ideal body weight (kg) = [height (cm) - 70] ´ 0.6 for female subjects
3. Acceptable medical history and physical examination including:

   * no particular clinically significant abnormalities in Electrocardiogram(ECG) results within six months prior to Period I dosing.
   * no particular clinical significance in general disease history within two months prior to Period I dosing.
4. Acceptable biochemistry determinations (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes ASpartate aminoTransferase (AST), ALanine aminoTransferase (ALT), Gamma-Glutamyl-Transpeptidase (g-GT), alkaline phosphatase, total bilirubin, albumin, glucose, BUN, uric acid, creatinine, total cholesterol, and triglyceride (TG).
5. Acceptable hematology (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes hemoglobin, hematocrit, red blood cell count, white blood cell count with differentials and platelets.
6. Acceptable urinalysis (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes pH, blood, glucose, ketones, bilirubin and protein.
7. Female of childbearing potential practicing an acceptable method of birth control for the duration of the study.
8. Have signed the written informed consent to participate in this study.

Exclusion Criteria:

1. A clinically significant disorder involving the cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the investigator).
2. A clinically significant illness or surgery within four weeks prior to Period I dosing (as determined by the investigator).
3. History of gastrointestinal obstruction, inflammatory bowel disease, gallbladder disease, pancreas disorder over last two years or history of gastrointestinal tract surgery over last five years.
4. History of kidney disease or urination problem over last two years deemed by the investigator to be clinically significant.
5. Known or suspected history of drug abuse within lifetime as judged by the investigator.
6. History of alcohol addiction or abuse within last five years as judged by the investigator.
7. History of allergic response(s) to voriconazole, any other drugs analogous to voriconazole, or any antibiotics.
8. Evidence of chronic or acute infectious diseases.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2020-06-21 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | 0 (pre-dose), 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10, 12, 24, and 36 hours
  The 90% confidence intervals of the geometric mean ratio (test/reference) for all parameters of voriconazole should fall within the range of 80.00% and 125.00%.
Time to reach peak concentration (Tmax) | 0 (pre-dose), 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10, 12, 24, and 36 hours
  The 90% confidence intervals of the geometric mean ratio (test/reference) for all parameters of voriconazole should fall within the range of 80.00% and 125.00%.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC 0-t) | 0 (pre-dose), 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10, 12, 24, and 36 hours
  The 90% confidence intervals of the geometric mean ratio (test/reference) for all parameters of voriconazole should fall within the range of 80.00% and 125.00%.
Area under the plasma concentration-time curve from time zero to infinity (AUC 0-∞) | 0 (pre-dose), 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10, 12, 24, and 36 hours
  The 90% confidence intervals of the geometric mean ratio (test/reference) for all parameters of voriconazole should fall within the range of 80.00% and 125.00%.
Elimination rate constant (入z) | 0 (pre-dose), 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10, 12, 24, and 36 hours
  The 90% confidence intervals of the geometric mean ratio (test/reference) for all parameters of voriconazole should fall within the range of 80.00% and 125.00%.
Terminal elimination half-life (t 1/2) | 0 (pre-dose), 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10, 12, 24, and 36 hours
  The 90% confidence intervals of the geometric mean ratio (test/reference) for all parameters of voriconazole should fall within the range of 80.00% and 125.00%.
Ratio of AUC 0-t to AUC 0-∞ | 0 (pre-dose), 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10, 12, 24, and 36 hours
  The 90% confidence intervals of the geometric mean ratio (test/reference) for all parameters of voriconazole should fall within the range of 80.00% and 125.00%.

SECONDARY OUTCOMES:
Adverse events and incidences | 0 (pre-dose), 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10, 12, 24, and 36 hours
  Any symptom, sign or significant abnormal laboratory finding whether observed or reported during the course of the study will be reported as an adverse event (AE) whether or not it has causative relationship with the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan